CLINICAL TRIAL: NCT03650192
Title: INVSENSOR00027 Clinical Performance Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-19415
Record Dates: First submitted 2018-08-27; First posted 2018-08-28 (Actual); Results first posted 2021-01-29 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- INVSENSOR00027 Test group (Experimental): The subjects will be enrolled into the test group and will receive the INVSENSOR00027 investigational sensor.
  Interventions: Device: INVSENSOR00027

INTERVENTIONS:
Device: INVSENSOR00027 — Investigational, noninvasive sensor that will be placed on the subject's chest and/or back. INVSENSOR00027 measures signals regarding subject's movement and posture, heart rate, and respiratory rate.

SUMMARY:
This study assesses the investigational sensor's (INVSENSOR00027) performance for detection of subjects' position and posture in bed, along with heart rate and respiratory rate.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* Physical status of ASA I or II
* Subjects must be able to read and communicate in English
* Has signed all necessary related documents, e.g. written informed consent, volunteer payment form, confidentiality agreement
* Has completed Health Assessment Questionnaire and passed health assessment screening

Exclusion Criteria:

* Subject has any medical condition which in the judgment of the investigator, renders them inappropriate for participation in this study
* Inability to tolerate sitting still or minimal movement for at least 30 minutes
* Nursing female volunteers
* Excluded at the Principal Investigator's discretion
* Refusal to take the pregnancy test (for female subjects)
* Positive pregnancy test for female subjects of child bearing potential. This is done for the safety of this population.
* Refusal to shave hair (neck, chest) off areas where sensors will be applied (male subjects)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Alghazi, Principal Investigator — Masimo Corporation
Locations (1):
- Masimo Clinical Lab, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00027 Test Group
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | INVSENSOR00027 Test Group
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 38
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 11
  Asian or Pacific Islander | 4
  Caucasian | 18
  Hispanic | 4
  Native American | 1
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of INVSENSOR00027's Posture Change Detection
Description: For each subject's position detection, INVSENSOR00027 output will be compared against observer's notes at each turn of the subject. Correctly detected position changes will be marked as True Positive. Missed detections (if any) will be counted. The sensitivity of INVSENSOR00027's posture change detection will be computed as Sensitivity = True Positive/(True Positive+Missed Detection)
Time Frame: 1-5 hours
Measure: Number; unit: percent sensitivity for posture change
Arm/Group | INVSENSOR00027 Test Group
Number analyzed (Participants) | 40
percent sensitivity for posture change | 100

2. Primary Outcome: Sensitivity of INVSENSOR00027's Activity Change Detection
Description: For each subject's activity (e.g., walking and upright) detection, INVSENSOR00027 output will be compared against observer's notes. Correctly detected activity changes will be marked as True Positive. Missed detections (if any) will be counted. The sensitivity of INVSENSOR00027's activity change detection will be computed as Sensitivity = True Positive/(True Positive+Missed Detection).
Time Frame: 1-5 hours
Measure: Number; unit: percent sensitivity for posture change
Arm/Group | INVSENSOR00027 Test Group
Number analyzed (Participants) | 40
percent sensitivity for posture change | 96.7

3. Primary Outcome: Sensitivity of INVSENSOR00027's Fall Event Detection
Time Frame: 1-5 hours
Population: Fall detection was an optional event per protocol.
Measure: Number; unit: percent sensitivity for fall detection
Arm/Group | INVSENSOR00027 Test Group
Number analyzed (Participants) | 3
percent sensitivity for fall detection | 100

4. Secondary Outcome: Respiratory Rate Detection
Description: Accuracy will be determined by comparing the respiratory rate measurement of the INVSENSOR00027 to the respiratory rate reference (RRef) and calculating the arithmetic root mean square (Arms) value. In order to obtain the Arms value, the RR measurement from the reference is subtracted from the INVSENSOR00027 RR measurement for a number of samples. The average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms value.
Time Frame: 1-5 hours
Population: 2 subjects were excluded due to data collection issues.
Measure: Number; unit: A(RMS) of breaths per minute
Arm/Group | INVSENSOR00027 Test Group
Number analyzed (Participants) | 38
A(RMS) of breaths per minute | 1.7

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study (35 days).
Arm/Group | INVSENSOR00027 Test Group
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-07): https://cdn.clinicaltrials.gov/large-docs/92/NCT03650192/Prot_SAP_000.pdf